CLINICAL TRIAL: NCT03163160
Title: Intratissue Percutaneous Electrolysis Technique vs. Manual Therapy in Women With Dyspareunia and Pelvic Pain
Brief Title: Electrolysis Technique vs Manual Therapy in Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quirón Madrid University Hospital (Other)
Responsible Party: Principal Investigator, Carolina Walker Chao, PhD, Quirón Madrid University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BET116183
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Dyspareunia; Pelvic Pain; Pelvic Floor Disorders; Musculoskeletal Pain; Perineal Tear
Keywords: pelvic floor muscles; pelvic floor myalgia; manual therapy; electrolysis; galvanic
MeSH Terms: conditions — Dyspareunia; Pelvic Pain; Pelvic Floor Disorders; Musculoskeletal Pain; Vaginismus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor manual therapy group (Experimental): Pelvic floor manual therapy is a clinical approach utilizing specifics hands-on mobilizing techniques to treat soft tissues. The technique require mobilization of soft-tissue by myofascial stretching maneuvers intended to improve bio-mechanical elasticity. The therapeutic protocol will be applied for 4 weeks.
  Interventions: Procedure: Pelvic floor manual therapy group
- Pelvic floor electrolysis group (Experimental): Pelvic floor electrolysis technique consists in an ultrasound-guided application of a galvanic electrolytic current that causes a controlled local inflammatory process in the target tissue. This allows for phagocytosis and the subsequent regeneration of the affected tissue. The therapeutic protocol will be applied for 4 weeks.
  Interventions: Procedure: Pelvic floor electrolysis group

INTERVENTIONS:
Procedure: Pelvic floor manual therapy group — Soft-tissue (myofascial) stretching techniques on pelvic floor muscles through external and internal (intra-vaginal) mobilizations. One weekly session for four weeks.
  Other Names: Man Ther Group
  Arms: Pelvic floor manual therapy group
Procedure: Pelvic floor electrolysis group — An ultrasound-guided application of a galvanic electrolytic current with an acupuncture needle in the soft tissue of pelvic floor. EPI technique was applied using a specifically device (EPI-X Omega Advanced Medicine, Barcelona, Spain) which produces modulated galvanic electricity. This is applied using a modified electrosurgical scalpel that incorporates acupuncture needles (0.3 mm in diameter) of different lengths. The intensity can be adjusted by changing either the duration of stimulation or the output current (mA) of the device.
  One weekly session for four weeks.
  Other Names: EPI
  Arms: Pelvic floor electrolysis group

SUMMARY:
Pelvic floor muscle physical therapy is recommended in clinical guidelines for women dyspareunia and pelvic pain. This study compare pelvic floor manual therapy and intratissue percutaneous electrolysis (EPI) technique in the treatment of pelvic pain in women with dyspareunia. Half of participants will receive pelvic floor manual therapy while the other half will receive intratissue percutaneous electrolysis technique.

DETAILED DESCRIPTION:
Dyspareunia is painful sexual intercourse and causes could be related to musculoskeletal pelvic floor muscles disorders (tenderness, trigger points, scars). There is evidence that manual therapy and intratissue percutaneous electrolysis can be effective for musculoskeletal pain disorders affecting muscles, tendons and fascias of the extremities but they have not been evaluated in pelvic floor muscle pain syndrome. The aim of this study is to compare manual therapy and EPI in the treatment of pelvic pain in women with dyspareunia.

Pelvic floor manual therapy is a clinical approach utilizing specifics hands-on mobilizing techniques to treat soft tissues. Pelvic floor mobilization is a slow controlled process of soft-tissue (myofascial) stretching intended to improve bio-mechanical elasticity.

EPI technique consists in an ultrasound-guided application of a galvanic electrolytic current that causes a controlled local inflammatory process in the target tissue. This allows for phagocytosis and the subsequent regeneration of the affected tissue.

ELIGIBILITY:
Inclusion Criteria:

* women with pain in the perineal area at an average intensity of 5 or more on the Numerical Rating Scale (NRS) during penetration or during pelvic examination, which is indicative of moderate to severe pain
* At least three months postpartum or any gynecology surgery

Exclusion Criteria:

* pregnancy
* active urinary or vaginal infection
* pelvic pathology associated with a lower genital pain problem (e.g. deep dyspareunia) and constant, spontaneous vulvar pain
* younger than 18 or older than 65 years
* previous interventions with steroid injections
* fibromyalgia syndrome

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Pain intensity before and after the intervention | Seven days after weekly session
  Changes in pain intensity before and after the intervention. A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of perineal pain during the external and intra-vaginal examination.

SECONDARY OUTCOMES:
Female sexual function index | Seven days after the last session and three months later
  Sexual function measure by the six-item Female Sexual Function Index (FSFI-6)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Walker, PT, PhD, Principal Investigator — Hospital Universitario Quiron Madrid
Locations (1):
- Hospital Universitario Quirón Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Signorello LB, Harlow BL, Chekos AK, Repke JT. Postpartum sexual functioning and its relationship to perineal trauma: a retrospective cohort study of primiparous women. Am J Obstet Gynecol. 2001 Apr;184(5):881-8; discussion 888-90. doi: 10.1067/mob.2001.113855. PMID 11303195
- [Background] Leeman LM, Rogers RG. Sex after childbirth: postpartum sexual function. Obstet Gynecol. 2012 Mar;119(3):647-55. doi: 10.1097/AOG.0b013e3182479611. PMID 22353966
- [Background] Yong PJ, Mui J, Allaire C, Williams C. Pelvic floor tenderness in the etiology of superficial dyspareunia. J Obstet Gynaecol Can. 2014 Nov;36(11):1002-1009. doi: 10.1016/S1701-2163(15)30414-X. PMID 25574678
- [Background] Bedaiwy MA, Patterson B, Mahajan S. Prevalence of myofascial chronic pelvic pain and the effectiveness of pelvic floor physical therapy. J Reprod Med. 2013 Nov-Dec;58(11-12):504-10. PMID 24568045
- [Background] Zoorob D, South M, Karram M, Sroga J, Maxwell R, Shah A, Whiteside J. A pilot randomized trial of levator injections versus physical therapy for treatment of pelvic floor myalgia and sexual pain. Int Urogynecol J. 2015 Jun;26(6):845-52. doi: 10.1007/s00192-014-2606-4. Epub 2014 Dec 20. PMID 25527482
- [Background] Abat F, Gelber PE, Polidori F, Monllau JC, Sanchez-Ibanez JM. Clinical results after ultrasound-guided intratissue percutaneous electrolysis (EPI(R)) and eccentric exercise in the treatment of patellar tendinopathy. Knee Surg Sports Traumatol Arthrosc. 2015 Apr;23(4):1046-52. doi: 10.1007/s00167-014-2855-2. Epub 2014 Jan 30. PMID 24477495
- [Background] Moreno C, Mattiussi G, Nunez FJ, Messina G, Rejc E. Intratissue percutaneous electolysis combined with active physical therapy for the treatment of adductor longus enthesopathy-related groin pain: a randomized trial. J Sports Med Phys Fitness. 2017 Oct;57(10):1318-1329. doi: 10.23736/S0022-4707.16.06466-5. Epub 2017 Jan 23. PMID 28116876
- [Background] Mattiussi G, Moreno C. Treatment of proximal hamstring tendinopathy-related sciatic nerve entrapment: presentation of an ultrasound-guided "Intratissue Percutaneous Electrolysis" application. Muscles Ligaments Tendons J. 2016 Sep 17;6(2):248-252. doi: 10.11138/mltj/2016.6.2.248. eCollection 2016 Apr-Jun. PMID 27900300
- [Background] Arias-Buria JL, Truyols-Dominguez S, Valero-Alcaide R, Salom-Moreno J, Atin-Arratibel MA, Fernandez-de-Las-Penas C. Ultrasound-Guided Percutaneous Electrolysis and Eccentric Exercises for Subacromial Pain Syndrome: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:315219. doi: 10.1155/2015/315219. Epub 2015 Nov 15. PMID 26649058